CLINICAL TRIAL: NCT00984776
Title: Detection of Vulnerable Plaque With Coronary Vessel Wall MRI: Contrast Enhanced MRI With Gadofosveset MS-325.
Brief Title: Detection of Coronary Vulnerable Plaque With Contrast-enhanced Magnetic Resonance Imaging
Acronym: T9M
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Bayer (Industry)
Responsible Party: T. Leiner, M.D., PhD, Maastricht University Medical Center
Purpose: Diagnostic
Other Study IDs: MEC 06-1-036
Record Dates: First submitted 2009-09-23; First posted 2009-09-25 (Estimated); Last update posted 2009-09-25 (Estimated); Status verified 2009-09

CONDITIONS: Coronary Artery Disease; Stable Angina; Unstable Angina
Keywords: coronary artery; MRI; vessel wall imaging
MeSH Terms: conditions — Coronary Artery Disease; Angina, Stable; Angina, Unstable | interventions — gadofosveset trisodium

INTERVENTIONS:
Other: Contrast enhanced MRI with Gadofosveset — 0.03 mmol/kg bodyweight of gadofosveset will only once be administered during MRI procedure via an intravenous catheter
  Other Names: Vasovist; MS-325

SUMMARY:
MRI has the ability to visualize the arterial vessel wall. Wall thickening and atherosclerotic plaque components can be visualized in the carotid arteries and the aorta. Previous studies also demonstrated the ability of MRI to visualize the coronary vessel wall. The ultimate goal of coronary vessel wall imaging is to detect vulnerable atherosclerotic plaque thereby. This might prevent complications, e.g., chest pain (angina) or myocardial infarction.

The goal of this study was to validate MRI of the coronary vessel wall by comparing it to intravascular ultrasound (IVUS), to detect atherosclerotic plaque in the coronary vessel wall and to look at the uptake of the albumin-binding contrast agent gadofosveset in atherosclerotic plaques. The main hypothesis is that due to the albumin binding characteristics, uptake of the contrast agent will take place in the more vulnerable plaques compared to less vulnerable plaques. MRI will be compared to X-ray coronary angiography and intravascular ultrasound, two techniques currently considered as the standard of reference for imaging of the coronary arteries and vessel wall.

ELIGIBILITY:
Inclusion Criteria:

* scheduled X-ray angiography for known coronary artery disease, valvular disease or chest pain with unknown origin
* age > 18 yrs and < 90 yrs
* Informed consent

Exclusion Criteria:

* arrhythmia
* hemodynamic unstable patients
* contra-indications for (contrast-enhanced) MRI
* age < 18 yrs or > 90 yrs

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-03; Primary Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Validation of MRI: comparison with IVUS. Can plaque be detected? | 1 week

SECONDARY OUTCOMES:
uptake contrast agent gadofosveset in atherosclerotic plaque in the coronary vessel wall? | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Tim Leiner, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands

REFERENCES:
- [Derived] Gerretsen S, Kessels AG, Nelemans PJ, Dijkstra J, Reiber JH, van der Geest RJ, Katoh M, Waltenberger J, van Engelshoven JM, Botnar RM, Kooi ME, Leiner T. Detection of coronary plaques using MR coronary vessel wall imaging: validation of findings with intravascular ultrasound. Eur Radiol. 2013 Jan;23(1):115-24. doi: 10.1007/s00330-012-2576-1. Epub 2012 Jul 11. PMID 22782568